CLINICAL TRIAL: NCT04936100
Title: Assessment of the Validity, Reliability, and Feasibility of Two Smartphone Applications for Testing the Visual Acuity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 99424
Record Dates: First submitted 2021-04-25; First posted 2021-06-23 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2021-04

CONDITIONS: Vision Impairment; Blindness
Keywords: Visual acuity; Smartphone
MeSH Terms: conditions — Vision Disorders; Blindness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Visual acuity assessment using "Vision Screening module" of "Easy Vision" application (Experimental)
  Interventions: Device: Assessment of distance and near visual acuity using "Vision Screening module" of "Easy Vision" application
- Visual acuity assessment using "Test Yourself module" of "Easy Vision" application (Experimental)
  Interventions: Device: Assessment of distance and near visual acuity using "Test Yourself module" of "Easy Vision" application
- Visual acuity assessment using "Peek Acuity" application (Experimental)
  Interventions: Device: Assessment of distance and near visual acuity using "Peek Acuity" application
- Visual acuity assessment using the conventional methods (Other)
  Interventions: Other: Assessment of distance and near visual acuity using the conventional methods

INTERVENTIONS:
Device: Assessment of distance and near visual acuity using "Vision Screening module" of "Easy Vision" application — The presenting visual acuity will be assessed using the Vision Screening module of the "Easy Vision" application.
  Arms: Visual acuity assessment using "Vision Screening module" of "Easy Vision" application
Device: Assessment of distance and near visual acuity using "Test Yourself module" of "Easy Vision" application — The presenting visual acuity will be assessed using the Test Yourself module of the "Easy Vision" application.
  Arms: Visual acuity assessment using "Test Yourself module" of "Easy Vision" application
Device: Assessment of distance and near visual acuity using "Peek Acuity" application — The presenting visual acuity will be assessed using the "Peek Acuity" application.
  Arms: Visual acuity assessment using "Peek Acuity" application
Other: Assessment of distance and near visual acuity using the conventional methods — The presenting visual acuity will be assessed using the conventional methods ["Chart: Tumbling E optotype" for assessing distance visual acuity and "Handheld chart: Tumbling E Near Point Vision Chart" for assessing near visual acuity]
  Arms: Visual acuity assessment using the conventional methods

SUMMARY:
Visual acuity (VA) is the most common measure of visual function globally. In clinical settings and during screening events, VA is an important measure to quantify changes in vision over time. Additionally, in the context of epidemiological studies and population-based surveys, VA is a critical measure to determine the presence and degree of vision impairment and to report on the indicators of effective eye care service coverage (i.e. refractive error and cataract surgery), that are currently considered by World Health Organization (WHO) for monitoring progress towards the Universal Health Coverage.

There are numerous applications for assessing VA; however, the number of validated applications is limited. In this study, the investigators aim to evaluate the external validity, intra- and inter-observer reliability, and feasibility of two applications ("Easy Vision" and "Peek Acuity") for testing the visual acuity.

ELIGIBILITY:
Inclusion criteria:

• Age ≥10 years old

Exclusion criteria:

• Subjects who are not able to respond to the examiner

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Distance visual acuity assessment with Easy Vision versus Peek Acuity versus conventional distance visual acuity chart | Through study completion [an average of 6 months]
  To assess the agreement between two smartphone-based evaluation of distance visual acuity (LogMAR unit) with Easy Vision and Peek Acuity and a conventional distance visual acuity chart (Tumbling E optotype)
Near visual acuity assessment with Easy Vision versus Peek Acuity versus conventional near visual acuity chart | Through study completion [an average of 6 months]
  To assess the agreement between two smartphone-based evaluation of near visual acuity (LogMAR unit) with Easy Vision and Peek Acuity and a conventional near visual acuity chart (Handheld chart: Tumbling E Near Point Vision Chart)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences, Tehran, Iran